CLINICAL TRIAL: NCT03684148
Title: Effects of Motor Imagery Intervention on Functional Recovery Following Total Knee Arthroplasty
Acronym: KSV2017
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Science and Research Centre Koper (Other)
Collaborators: Slovenian Research Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Knee Study Valdoltra 2017
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Osteo Arthritis Knee; Knee Arthroplasty
Keywords: osteoarthritis; muscle voluntary activation; knee replacement; cognitive training; functional performance; randomized controlled trial
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: This was a randomized, controlled, parallel-group intervention trial to evaluate the benefits of adding MI practice to CPT postoperative rehabilitation program. Eligible patients were randomly assigned to either an intervention group in which MI practice was combined with CPT (MIp), or to a control group which received CPT alone (CON).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor imagery practice (Experimental): In addition to routine physical therapy patients that will be included in the motor imagery practice (MIp) group will receive an additional intervention based on motor imagery beginning immediately after the TKA procedure.
  Interventions: Other: Motor imagery practice
- Control group (No Intervention): Patients from the control group will underwent the same post-surgery rehabilitation program, but will not be engaged in MI practice.

INTERVENTIONS:
Other: Motor imagery practice — In detail, they were advised to imagine maximal voluntary isometric contractions (MViC). MViC imagery practice was planned in a progressive manner. Thus, it was performed in two sets of 25 repetitions with 2 minutes of inter-sets rest period, for two weeks, and 10 additional repetitions were added on week three and four, respectively. Each MViC repetition was sustained for 5 seconds, followed by 5 seconds of inter-repetition rest periods. Additionally, after every fifth contraction, participants had a 20 seconds of rest. Following 5 days of MI practice, the participants were advised to take a break from MI for two consecutive days. After hospital discharge, the participants in the MIp group were supplied with an audio description of the exercises to be performed.
  Other Names: Routine physical therapy
  Arms: Motor imagery practice

SUMMARY:
The knee osteoarthritis becoming a leading cause of disability among older adults' population. When conventional treatments fail, a total knee arthroplasty (TKA) is suggested. Although TKA treatment significantly reduces pain and improve mobility of patients, there is still high prevalence of patients whose neuromuscular function is impaired up to three years following TKA, which can be directly prescribed to poor or/and inadequate rehabilitation practice. Thus, motor imagery (MI) is proposed as additional rehabilitation tool to convention physical therapy to reduce decline of neuromuscular function in early days post-surgery. Recent studies showed that MI could facilitate learning and acquisition of motor skills, as well as maintain and retain previously acquired motor skills, which may be beneficial for those who undergo TKA. It represents an incentive in the process of motor learning and the transfer of the mental scheme of the motion pattern into the process of movement execution. Measuring neuromuscular function pre- and post-TKA could be unique opportunity to provide empirical evidence about its additional therapeutic effects. Outcomes of proposed research project could serve to improve existing intervention programs applied in rehabilitation protocols following TKA surgery as well as other orthopedic interventions. This would also contribute to the successful return of individuals after an injury to their everyday working routine. We hypothesized that MI practice group will experience better both subjective and objective measures of functional performance compared to control group that will be subjected to routine physical therapy only.

DETAILED DESCRIPTION:
TKA is widely considered to have a successful outcomes, comparing pre and postoperative scores on pain and both subjective and objective functional measures. Nevertheless, a significant proportion of patients report continuing pain, functional limitations, and dissatisfaction up to three years after the surgery. Thus we planed to conduct intervention study.

OBJECTIVES:

• Primary goal of the research is to determine how the MI practice intervention will influences on the recovery of neuromuscular and locomotor function following TKA.

Specific goals of the research are as follows:

* To examine effects of MI practice intervention to other measured parameters as follows:

  1. maximal isometric strength of knee extensors,
  2. maximal voluntary activation level
  3. spatio-temporal gait parameters during different gait velocities under single- and dual-task conditions,
  4. contractile muscle parameters,
  5. electromechanical efficiency index,
  6. self-reported measure of knee function (OKS and LEFS),
  7. and pain level assessed by Visual Analogue Scale (VAS).

     HYPOTHESIS:

     The main hypothesis of this dissertation is that the group, which will perform motor imagery practice intervention will have fewer decline in motor functions following TKA surgery.

     H1: Motor imagery (MI) leads to lower functional decline at one-month period after surgery as compared to control group (CON).

     H1.1: Patients in MI intervention group have fewer decline in maximal isometric knee extensors strength.

     H1.2: Patients in MIp intervention group have fewer decline in spatio-temporal gait parameters during different gait velocities under single- and dual-task conditions.

     H1.3: Patients in MI intervention group have fewer decline in voluntary muscle activation level.

     H1.4: Patients in MI intervention group will not experience significantly greater decline in contractile muscle parameters as compared to CON group.

     H1.5: Patients in MI intervention group have fewer decline in electromechanical efficiency index.

     H1.6: Patients in MI intervention group have better self-reported knee function assessed by self-reported questionnaires.

     H1.7: Patients in MI intervention group have fewer pain level assessed by VAS.
     1. Methods

     Participants:

     N = 26 (man/woman) of which:

  <!-- -->

  1. Symptomatic population / n = 26; have already determined date for TKA surgery

     Participants will be recruited from Valdoltra orthopedic hospital (Ankaran, Slovenia).

     Inclusion criteria: scheduled for unilateral TKA secondary to osteoarthritis; age from 50 to 80 years old; participants were not engaged in preoperative treatments;

     Exclusion criteria: participants who had a previous history of TKA on the same side as the surgery; body mass index of 40 kg/m2 or higher; bilateral TKA's; patients with a history of any neurological disorder including Cerebral Vascular Attack, Multiple Sclerosis, or Parkinson's disease; patients with Rheumatoid Arthritis or active cancer; thrombose; bleeding after surgery; previously participation in imagery training.

     Sample Size:

     Isometric knee extension strength of the surgical leg was defined as the primary outcome variable for the power analysis. The sample size was calculated based on Hopkins recommendations (W. G. Hopkins, 2006) using online available spreadsheet (http://sportsci.org/resource/stats/index.html). Raw mean difference in change (RDC) was calculated based on pilot study of my own (RDC = 48,51 Nm) (unpublished data). Further, minimal clinically important change (MCIC) (MCIC = 21,89 Nm) (van der Roer, Ostelo, Bekkering, van Tulder, & de Vet, 2006) was calculated based on standard error of measurement (SEM) (SEM = 7,9 Nm) from study of Lienhard (Lienhard et al., 2013) that assessed reliability of isometric knee extensor strength of TKA patients. Given that in clinical practice the drop out of subjects is common because of many reasons (aging process, comorbidities, post-surgery complications), we adjusted originally calculated sample size by following formula: N1 = n/(1-d) (Sakpal, 2010) where N1 is adjusted sample size, n is the sample size required as per proposed formula ( N = 7 per group) and d is the drop-out rate (d = 0,25). This resulted in a target sample size of 10 in each of two groups (Mip and control). The recruitment of the patients will continue until the target sample size is achieved.

     2. Procedure

     - Ethical permission (already approved) - Ethics Committee of Valdoltra orthopedic hospital.

     - Measurement assessment participants PRE-surgery (one day before surgery on average)

     - MI practice intervention

     - Measurement assessment participants POST-surgery 1 (one month after surgery on average)

     - Measurement assessment participants POST-surgery 2 (one year after surgery on average)

     The patients will be randomized into two groups: the experimental MI practice group (MIp) and control group (CON), which will have common in patient and home-based physical therapy only. Subjects in both groups will receive one daily continuous passive motion (CPM) session (Kinetec Performa), beginning on the second day after TKA (immediately after intensive care) until discharge (5 to 7 days). Nurses will install the CPM device, by the standardized procedure. Identical installations will be performed for both groups: subjects laying supine in their bed, and the CPM device will be placed under the operated leg with the knee extended. For stability, one strap will surround the subject's thigh, another strap surrounds the subject's lower leg, and the apparatus will be prevented from sliding down by the edge of the bed. The CPM will be used for 45 minutes continuously, including a 5-minute warm-up period.

     Patients included in MI group will have intervention based on motor imagery technique with beginning immediately after intensive care. In detailed, they will be advised to imagine maximal voluntary isometric contractions (MViC). MViC imagery practice will be progressive. Thus, it will be performed in two sets of 25 repetitions with 2 minutes of inter-sets rest period, with 10 additional trials in week three and four. Each MViC repetition should be sustained for 5 seconds, followed by 5 seconds of inter-repetition rest periods. Additionally, after every five contractions, participants will have a 20 seconds of rest in order to minimize the onset of mental fatigue (Rozand, Lebon, Stapley, Papaxanthis, & Lepers, 2016). Following 5 days of MIp the participants were advised to take a break from MIp for two days in a raw.

     After release from the hospital participants from MIp group will be supplied with audio description of exercise they need to perform in order to better concentrate to MIp task, rather than programme variables itself. Additionally, after release from hospital both groups will be supplied with a physical exercise program that they need to perform in home-based environment (like that one they will have in the hospital). In general, exercise programme considered active and passive knee flexion, abduction and adduction of the hip in the horizontal plane. Knee extensor muscle strengthening exercises such as unilateral knee extension with resistance of healthy leg, bilateral sit up from the higher chair/the high was adjusted by the pillow, unilateral weight bearing eccentric contraction supported with crutches etc. Next, functional exercises with weight bearing were adviced with attention of transferring the preasure (personal weight) on operated leg as much as possible.

     Each participant will be called by the phone every day in order to monitor their adherence to the prescribed exercise programme (lower than 80% of adherence will be excluded from the post analysis).

     Given that reported placebo effect in psychological outcomes of exercise training is small (ES = 0,20) (Lindheimer, O'Connor, & Dishman, 2015), to control it and additional socio-psychological influence of MIp instructor on the MIp outcomes, we will ensure the same conditions for the other group and spend the same amount of time with them (approximately 15 minutes per day) with each patient (verbal communication on site/in hospital or by telephone call/after discharge) regardless of his randomization to the group.

     Measurement assessments:

     Measurement assessment will be conducted in period before TKA (BT), and 1 month after the surgery.We will evaluate:

     I. Cognitive assessment:

     - Montreal Cognitive Assessment (MoCA): cognitive screening tool for Mild Cognitive Impairment

     II. Anthropometry:

     - Body weight and height (Stable stadiometer Seca, Birmingham, UK) and body composition (Bio-impedance system MALTRON BF-906).

     III. Functional status:

     - flexibility of knee joint (flexion and extension ROM) - assessed by manual goniometer

     - agility and dynamic balance (Timed "Up & Go" Test)

     - Sit to stand (30 seconds)

     - spatio-temporal gait parameters (STGP) during different gait velocities will be measured by OPTOGAIT system (Microgate, Bolzano, Italy) under single- and dual-task conditions.
     * Hand grip strength along with both the knee extensors and flexors muscles maximal voluntary isometric strength (MViC) (isometric dynamometer S2P)
     * Self - reported functional assessment (OKS and LEFS questionnaires)

     IV. Muscle function:
     * contractile muscle parameters (Tensiomyography)
     * electromechanical efficiency index (Tensiomyography and M-wave module)
     * Voluntary activation level (using double interpolated twitch technique) V. Pain level - Visual analogue scale (VAS)

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for unilateral TKA secondary to osteoarthritis;
* age from 50 to 80 years old;
* participants were not engaged in preoperative treatments

Exclusion Criteria:

* participants who were undergoing a revision TKA;
* body mass index (BMI) greater than 40 kg/m2;
* participants who were receiving a bilateral TKA's;
* uncontrolled hypertension;
* diabetes mellitus;
* a history of any neurological disorder;
* multiple sclerosis;
* Parkinson's disease;
* patients with rheumatoid arthritis or active cancer;
* previous history of deep vein thrombosis;
* contralateral knee OA (as defined by pain greater than 4/10 with activity)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Change in maximal voluntary isometric contraction of quadriceps muscle following a total knee arthroplasty | At baseline (1 day before surgery) and one month postoperatively
  Maximal strength assessed by isometric dynamometer

SECONDARY OUTCOMES:
Change in quadriceps muscle voluntary activation following a total knee arthroplasty | At baseline (1 day before surgery) and one month postoperatively
  Voluntary activation level was assessed by double interpolated twitch technique
Change in range of motion of knee joint following a total knee arthroplasty | At baseline (1 day before surgery) and one month postoperatively
  Flexion and extension range of motion of knee joint, assessed by manual long-arm goniometer
Change in agility following a total knee arthroplasty | At baseline (1 day before surgery) and one month and one year postoperatively
  Agility and dynamic balance will be assessed by timed up to go test
Change in repetitive strength of knee extensor muscles following a total knee arthroplasty | At baseline (1 day before surgery) and one month postoperatively and one year postoperatively
  Repetitive strength of knee extensor muscles will be assessed by chair sit to stand test
Change in spatio temporal gait parameters following a total knee arthroplasty | At baseline (1 day before surgery) and one month postoperatively
  Spatio-temporal gait parameters (STGP) during different gait velocities will be measured by OPTOGAIT system (Microgate, Bolzano, Italy) under single- and dual-task conditions
Change in hand grip strength following a total knee arthroplasty | At baseline (1 day before surgery) and one month postoperatively and one year postoperatively
  Hand grip strength will be measured by hand held dynamometer
Change in functional assessment scale measured by Oxford Knee Score following a total knee arthroplasty | At baseline (1 day before surgery) and one month postoperatively and one year postoperatively
  Self - reported functional assessment was measured by Oxford Knee Score (OKS) questionnaire. The OKS is a 12-item patient-reported PRO specifically designed and developed to assess function and pain after total knee arthroplasty (TKA) surgery. Each item can be scored from 1 to 5 points depending on patients pain and/or functional status level. Greater the score, better is function. It is short, reproducible, valid and sensitive to clinically important changes.
Change in functional assessment scale measured by Lower Extremity Functional Scale following a total knee arthroplasty | At baseline (1 day before surgery) and one month postoperatively and one year postoperatively
  Self - reported functional assessment was measured by Lower Extremity Functional Scale (LEFS). That is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress and outcome, as well as to set functional goals.
  The LEFS can be used to evaluate the functional impairment of a patient with a disorder of one or both lower extremities. It can be used to monitor the patient over time and to evaluate the effectiveness of an intervention. The columns on the scale are summed to get a total score. The maximum score is 80. The greater the score, function is better.
Change in contractile muscle parameters following a total knee arthroplasty | Participants will be assessed 1 day before surgery and one month postoperatively
  Contractile muscle parameters will be assessed by Tensiomiography (TMG). TMG will be used to detect muscle belly enlargement in transversal plane during an isometric twitch contraction with a means of digital high-precision displacement sensor. From TMG following parameters will be derived:
  Time of contraction (Tc) Sustain time (Ts) Relaxation time (Tr) Delay time (Td) and Displacement of muscle belly (Dm)
Change in electromechanical efficiency index following a total knee arthroplasty | At baseline (1 day before surgery) and one month postoperatively
  Electromechanical efficiency index will be assessed by Tensiomyography and M-wave module
Change in self perceived pain level following a total knee arthroplasty | At baseline (1 day before surgery) and one month postoperatively and one year postoperatively
  Self perceived pain level will be assessed by Visual Analog Scale (VAS). The VAS is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points from 1 to 100. Greater the score, greater the level of self perceived level of pain of patient.

CONTACTS AND LOCATIONS:
Overall Officials: Rado Pisot, PhD, Study Director — Science and Research Centre Koper
Locations (1):
- Orthopaedic Hospital Valdoltra, Ankaran, Slovenia

IPD SHARING:
Plan to Share IPD: No
We are willing to share supplementary material such as study protocol, measurement assessment protocol, motor imagery script used in intervention etc.

REFERENCES:
- [Result] Paravlic AH, Pisot R, Marusic U. Specific and general adaptations following motor imagery practice focused on muscle strength in total knee arthroplasty rehabilitation: A randomized controlled trial. PLoS One. 2019 Aug 14;14(8):e0221089. doi: 10.1371/journal.pone.0221089. eCollection 2019. PMID 31412056
- [Derived] Paravlic AH, Maffulli N, Kovac S, Pisot R. Home-based motor imagery intervention improves functional performance following total knee arthroplasty in the short term: a randomized controlled trial. J Orthop Surg Res. 2020 Oct 2;15(1):451. doi: 10.1186/s13018-020-01964-4. PMID 33008432
- See also: Online article — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0221089